CLINICAL TRIAL: NCT06605287
Title: A Study to Observe the Progress of Diabetes After Supaglutide Injection for 52 or 28 Weeks Treatment in Type 2 Diabetes Patients
Brief Title: The Progress of Diabetes After Supaglutide Treatment in Type 2 Diabetes Patients
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20230310-07
Record Dates: First submitted 2023-05-03; First posted 2024-09-20 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: clinical remission; Supaglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collect serum samples for cytokine detection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Supaglutide Treatment: Type 2 diabetes patients without any hypoglycemic drugs after 52 or 28 weeks of Supaglutide treatment

SUMMARY:
Glucagon like peptide-1 receptor agonist (GLP-1RA) can enhance insulin secretion and inhibit glucagon secretion in a glucose concentration dependent manner, delay gastric emptying, and reduce food intake through central appetite inhibition, thus achieving the effect of lowering glucose. Supaglutide Injection (YN-011, Diabegone®) has the characteristic of high affinity with GLP-1 receptors. Previous studies by Weng Jianping had shown that early use of short-term insulin fortification and oral medication (sulfonylureas and metformin) fortification therapy for newly diagnosed T2DM still resulted in clinical remission in about 50% of patients one year after discontinuation of medication, i.e. no hypoglycemic drugs were used, only diet and exercise therapy were maintained. At the same time, early fortification therapy can promote pancreatic islets β Cell repair. At present, there are few studies on the clinical remission rate of diabetes after GLP-1RA hypoglycemic treatment for one year. This study aims to discontinue the use of Supaglutide treatment after 52 or 28 weeks, and continue a one-year non pharmacological intervention observation to observe the clinical remission rate of diabetes, the changes in pancreatic islets β and α cell function, insulin resistance, body composition, and blood glucose fluctuations of patients who stopped using Supaglutide for 3 months and 1 year .

DETAILED DESCRIPTION:
With the rapid development of economy, the occurrence of diabetes in China has also shown a momentum of rapid growth. Dietary control and exercise are usually the foundation for treating T2DM. For patients whose glucose control does not meet the standard, hypoglycemic drugs should be added on the basis of diet control and exercise. Glucagon like peptide-1 receptor agonist (GLP-1RA) can enhance insulin secretion and inhibit glucagon secretion in a glucose concentration dependent manner, delay gastric emptying, and reduce food intake through central appetite inhibition, thus achieving the effect of lowering glucose. Supaglutide Injection (YN-011, Diabegone®) has the characteristic of high affinity with GLP-1 receptors. Supaglutide can activate GLP-1 receptor in pancreatic islets β cells to increase insulin secretion and inhibit glucagon release in a glucose dependent manner. Previous studies by Weng Jianping had shown that early use of short-term insulin fortification and oral medication (sulfonylureas and metformin) fortification therapy for newly diagnosed T2DM still resulted in clinical remission in about 50% of patients one year after discontinuation of medication, i.e. no hypoglycemic drugs were used, only diet and exercise therapy were maintained. At the same time, early fortification therapy can promote pancreatic islets β Cell repair. At present, there are few studies on the clinical remission rate of diabetes after GLP-1RA hypoglycemic treatment for one year. This study aims to discontinue the use of Supaglutide treatment after 52 or 28 weeks, and continue a one-year non pharmacological intervention observation to observe the clinical remission rate of diabetes, pancreatic islets β and α cell function, insulin resistance, changes in body composition, and blood glucose fluctuations of patients who stopped using Supaglutide for 3 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Complete a multicenter, randomized, double-blind, placebo-controlled clinical study on the efficacy of Supaglutide in T2DM patients with poor glucose control after dietary and exercise interventions (YN011-301);
* HbA1c ≤ 7.0%;
* The researchers determined that the patient's glucose control was stable based on the visit data of the subjects during the treatment with Supaglutide and the testing indicators of our hospital;
* The subjects agree to maintain scientific dietary and exercise habits throughout the entire research process, regularly conduct SMBG and keep records;
* Able to understand and willing to sign a written informed consent form and comply with the research protocol.

Exclusion Criteria:

* The researchers believe that the subjects have a disease state where they cannot complete the observation period follow-up;
* The researchers determined that there were situations in the subjects that affected the compliance of this study during the treatment with Supaglutide.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study, subjects with type 2 diabetes treated with Supaglutide were screened to meet the target of glucose control when they completed 52 or 28 weeks of Supaglutide treatment respectively.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The clinical remission rate of diabetes | 48 weeks
  Concentration of HbA1c changes in type 2 diabetes patients without any hypoglycemic drugs for 48 weeks after Supaglutide treatment

SECONDARY OUTCOMES:
Concentration of MBG (mmol/L) changes | 48 weeks
  Concentration of MBG changes in type 2 diabetes patients without any hypoglycemic drugs for 48 weeks after Supaglutide treatment by FGM
hange in TIR(%), TAR(%), TBR(%) | 48 weeks
  TIR, TAR, TBR analysis in type 2 diabetes patients without any hypoglycemic drugs for 48 weeks after Supaglutide treatment by FGM
Change in MAGE | 48 weeks
  MAGE analysis in type 2 diabetes patients without any hypoglycemic drugs for 48 weeks after Supaglutide treatment by FGM
Change in CV | 48 weeks
  CV analysis in type 2 diabetes patients without any hypoglycemic drugs for 48 weeks after Supaglutide treatment by FGM
Concentration of FBG(mmol/L), PBG(mmol/L) changes | 48 weeks
  Concentration of FBG, PBG changes in type 2 diabetes patients without any hypoglycemic drugs for 48 weeks after Supaglutide treatment
Concentration of C-peptide(ng/ml) changes | 48 weeks
  Concentration of C-peptide changes in type 2 diabetes patients without any hypoglycemic drugs for 48 weeks after Supaglutide treatment
Concentration of Insulin (mU/L) changes | 48 weeks
  Concentration of Insulin changes in type 2 diabetes patients without any hypoglycemic drugs for 48 weeks after Supaglutide treatment
Concentration of glucagon (pmol/L) changes | 48 weeks
  Concentration of glucagon changes in type 2 diabetes patients without any hypoglycemic drugs for 48 weeks after Supaglutide treatment
Change in HOMA-IR | 48 weeks
  HOMA-IR analysis in type 2 diabetes patients without any hypoglycemic drugs for 48 weeks after Supaglutide treatment
Change in body composition (%) | 48 weeks
  Body composition analysis in type 2 diabetes patients without any hypoglycemic drugs for 48 weeks after Supaglutide treatment
Change in Dex bone density (T value) | 48 weeks
  Dex bone density analysis in type 2 diabetes patients without any hypoglycemic drugs for 48 weeks after Supaglutide treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jianhua Ma, Principal Investigator — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing Medical Univesity, Nanjing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sun R, Wang K, Yuan G, Shi B, Wang X, Shao A, Xu Y, Wang Q, Ma J. Diabetes Remission in Drug-Naive Patients with Type 2 Diabetes After Efsubaglutide Alfa Treatment. Adv Ther. 2026 Jan 7. doi: 10.1007/s12325-025-03467-2. Online ahead of print. PMID 41498879